CLINICAL TRIAL: NCT02582203
Title: Clinical and Economic Outcomes of Ceftaroline Fosamil for the Treatment of Acute Bacterial Skin and Skin Structure Infections Documented or at Risk of Methicillin-Resistant S. Aureus
Brief Title: Clinical and Economic Outcomes of Ceftaroline Fosamil for ABSSSI Documented or at Risk of MRSA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wayne State University (Other)
Collaborators: Henry Ford Hospital (Other); St. John Providence Health System (Other); Detroit Medical Center (Other); Forest Laboratories (Industry)
Responsible Party: Principal Investigator, Michael J. Rybak, Director, Anti-Infective Research Laboratory, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1111010324
Record Dates: First submitted 2015-10-16; First posted 2015-10-21 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Skin Diseases, Infectious; Staphylococcal Skin Infections
Keywords: Ceftaroline fosamil; Vancomycin; Acute bacterial skin and skin structure infections; Methicillin-resistant S. aureus
MeSH Terms: conditions — Skin Diseases, Infectious; Staphylococcal Skin Infections | interventions — Ceftaroline; Vancomycin

ARMS (2):
- Ceftaroline (Active Comparator): 600 mg IV (over 1 hour) every 12 hours for renal function > 50 mL/min, adjusted for renal function based on package insert for no more than 14 days.
  Interventions: Drug: Ceftaroline
- Vancomycin (Active Comparator): Dosed by institutional pharmacy protocol to reach goal trough level of 10 - 20 mg/L steady state concentration for no more than 14 days.
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: Ceftaroline
  Arms: Ceftaroline
Drug: Vancomycin
  Arms: Vancomycin

SUMMARY:
The proposed study is a prospective, open-label, randomized, multi-center trial of ceftaroline versus vancomycin for the treatment of ABSSSI in patients documented or at risk for MRSA. Patients admitted to the Detroit Medical Center, Henry Ford Hospital, or St. John Medical Center in Detroit Michigan with a documented ABSSSI between April 2012 and November 2015 will be evaluated for inclusion. Patients must present with at least 3 of the following local signs/symptoms: pain, tenderness, swelling erythema, warmth, drainage/discharge, induration, and lymph node swelling/tenderness. Patients will be randomized 1:1 ceftaroline or vancomycin with optional anaerobic and/or Gram-negative coverage. The assignment of study drug will follow a randomized list that was previously generated via a computerized random mix block generator (nQuery Advisor® 7.0) and available at each of the study sites. Patients will be randomized to ceftaroline intravenously at 600 mg infused over 1 hour every 12 hours for patients with normal renal function. Patients randomized to vancomycin will receive the standard 15 mg/kg dose based on total body weight infused over 1 hour q 12 hour, dose and interval adjusted based on creatinine clearance and via institution-specific pharmacy protocol to target serum trough concentrations of 10-20 mg/L within the first 72 hours. Outcomes measured in the Clinically Evaluable patient population include day two or three size reduction (percentage) and clinical response at end of therapy or discharge.

ELIGIBILITY:
Inclusion Criteria:

* Acute bacterial skin and skin structure infection (cellulitis, major abscess, surgical site infection)
* Presence of MRSA or documented risk factors for MRSA (prior antibiotic use 60 days, prior hospital exposure 180 days, skin ulcers, central venous catheter)
* Anticipating no less than two days of hospital admission
* Signed informed consent

Exclusion Criteria:

* Gas gangrene/progressive necrotizing infections
* Osteomyelitis
* Infections due to Gram-negative pathogens or other Gram-positive pathogens if S. aureus or Streptococcus is not present
* Pathogens known at the study entry to be resistant to ceftaroline or vancomycin
* Anticipated to require non-study antibiotic active against S. aureus for another reason
* Treatment for the current episode of ABSSSI for > 24 hours with another intravenous anti-MRSA antibiotic
* Surgical (I & D) as definitive/curative treatment
* Presence of prosthetic hardware or invasive devices suspected to be the source of infection but cannot be removed
* Life expectancy < 2 months
* Open burn wound > 30% total body surface area
* Pregnant or nursing mothers
* Known allergic reaction to vancomycin or ceftaroline

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2012-02; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Early Clinical Response | 48 to 72 hours after initiation of study drug
  Reduction of lesion size from baseline of at least 20%

SECONDARY OUTCOMES:
Overall Clinical Response | End or therapy or patient discharge [Up to 60 days]
  Cure: pretreatment signs and symptoms are improved or resolved and no additional antibiotic therapy is necessary
  * Improved: pretreatment signs and symptoms are improved and additional antibiotic therapy is necessary
  * Failure: Persistent, worsening, or new/recurrent signs and symptoms, antibiotics needed > 14 days, or the need for a change in antibiotic therapy
Length of stay | During hospitalization [Up to 60 days]
  Total duration of hospitalization

OTHER OUTCOMES:
Adverse Events | During treatment with study drug [Up to 60 days]
  Any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not related to the medicinal product.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Rybak, PharmD, MPH, Principal Investigator — Wayne State University
Locations (3):
- United States (3):
  - Detroit Medical Center, Detroit, Michigan
  - St. John Hospital and Medical Center, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan

REFERENCES:
- [Derived] Claeys KC, Zasowski EJ, Trinh TD, Casapao AM, Pogue JM, Bhatia N, Mynatt RP, Wilson SS, Arthur C, Welch R, Sherwin R, Hafeez W, Levine DP, Kaye KS, Delgado G, Giuliano CA, Takla R, Rieck C, Johnson LB, Murray KP, Gordon J, Reyes K, Hartman P, Davis SL, Rybak MJ. Open-Label Randomized Trial of Early Clinical Outcomes of Ceftaroline Fosamil Versus Vancomycin for the Treatment of Acute Bacterial Skin and Skin Structure Infections at Risk of Methicillin-Resistant Staphylococcus aureus. Infect Dis Ther. 2019 Jun;8(2):199-208. doi: 10.1007/s40121-019-0242-5. Epub 2019 Mar 27. PMID 30915685